CLINICAL TRIAL: NCT05953116
Title: Managing the Nutritional Needs of Older Filipino With Due Attention to Protein Nutrition and Functional Health (ManoPo) Study
Brief Title: Managing the Nutritional Needs of Older Filipino With Due Attention to Protein Nutrition and Functional Health Study
Acronym: ManoPo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Nutrition Research Institute, Philippines (Other Government)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Robby Carlo A. Tan, Senior Science Research Specialist, Food and Nutrition Research Institute, Philippines
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FIERC-2022-019
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Body Composition; Protein; Exercise; Functional Status
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The trial participants and researchers will be blinded during the conduct of the 12-week intervention. An independent third party will handle randomization and allocation of participants to either intervention group (DOST-FNRI protein drink + physical activity) or placebo group (placebo product + physical activity), while trying to ensure a balanced sex distribution between the groups.
  The intervention group will receive a protein-containing product which shall meet the target of 30g of protein per day of supplementation. Meanwhile, the placebo group will receive an isocaloric product (similar caloric value but with minimal to no protein content). Both products will have similar packaging, appearance, taste, and flavoring. A unique serial number only known by the independent third party will be used to differentiate between the two products. Unblinding of trial participants will be done after data analysis of a locked dataset.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): A protein product (combination of whey protein and plant-derived protein) in powdered form with flavoring. Product will be added to 180-200 mL of warm water prior to consumption.
  Interventions: Dietary Supplement: Nutrition supplementation; Other: Exercise
- Placebo Group (Placebo Comparator): An isocaloric product (made with maltodextrin) in powdered form with flavoring. Product will be added to 180-200 mL of warm water prior to consumption.
  Interventions: Dietary Supplement: Nutrition supplementation; Other: Exercise

INTERVENTIONS:
Dietary Supplement: Nutrition supplementation — Blinded researchers will provide the randomly assigned supplement product to the trial participants for a period of 90 days. Used packaging will be collected at the end of every week from each trial participant to monitor compliance.
  Other Names: Protein drink
Other: Exercise — Trained researchers will facilitate resistance-based exercises two to three times a week in an enclosed venue (gym). Trial participants will be assessed at baseline for one repetition maximum (1RM) which will serve as a basis for load progression. A target of 3 sets and 6-15 repetitions with at least 30 seconds rest in between sets will be performed by the trial participants under supervision of a trained researcher.
  Other Names: Resistance and group exercise

SUMMARY:
The study aims to determine the effect of protein nutrition and exercise on the body composition and functional capacity of Filipino older adults.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of nutrition supplementation and exercise intervention on the main indicators of sarcopenia in older adults such as body composition (fat mass and lean mass), muscle strength (leg and handgrip), and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Pre-sarcopenia/pre-frail
* Aged 60 years old and above, male or female
* Free-living in the community, ambulatory
* Able to respond to food recall/interview as self-declared
* Normal cardiac function as measured by resting ECG

Exclusion Criteria:

* Bed ridden, unable to perform exercise independently
* Presence of serious medical condition (i.e. cancer, existing fracture)
* Presence of unmanaged hypertension and/or type 2 diabetes or upon assessment of physician
* Renal Problem
* Under controlled or medically-supervised diet not flexible to include the intervention agent
* Allergic to any ingredients in the nutrition supplementation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass, as measured by dual-energy x-ray absorptiometry (DXA) | Baseline, Midline (6 weeks), Endline (12 weeks)
  Measurement of appendicular skeletal muscle mass index (ASMI) by dividing total muscle mass (kg) of appendages with height in meters squared
Change in muscle strength, as measured by grip strength and leg strength (Jamar, MicroFET) | Baseline, Midline (6 weeks), Endline (12 weeks)
  Handgrip strength is measured using a hydraulic hand dynamometer through maximum exertion of grip force (in kilograms).
  Leg strength is measured using a hand-held dynamometer. Participant will use strongest leg force to push against the resistance brought upon by the researcher while holding the measuring device.
Change in physical performance, as measured by timed up-and-go test | Baseline, Midline (6 weeks), Endline (12 weeks)
  Faster time duration to complete the test indicate lesser risk for falls
Change in physical performance, as measured by short physical performance battery | Baseline, Midline (6 weeks), Endline (12 weeks)
  Score ranges from 0 to 12 with a higher score indicating better functionality
Change in physical performance, as measured by 10-meter walk test | Baseline, Midline (6 weeks), Endline (12 weeks)
  Faster walking speed (in meters per second) indicate better functionality

CONTACTS AND LOCATIONS:
Overall Officials: Robby Carlo A Tan, Msc, Principal Investigator — Department of Science and Technology-Food and Nutrition Research Institute (DOST-FNRI)
Locations (1):
- Department of Science and Technology-Food and Nutrition Research Institute, City of Taguig, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No